CLINICAL TRIAL: NCT05318781
Title: Understanding the Impact of Radical Changes in Diet and the Microbiome on Brain Function and Structure: the EMBRACE Study
Brief Title: Impacts of Bariatric Surgery on the Microbiome and Brain Function
Acronym: EMBRACE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Collaborators: Concordia University, Montreal (Other); Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other); University of Ottawa (Other)
Responsible Party: Principal Investigator, Simon Bacon, Professor, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Other Study IDs: MP-32-2022-2412
Record Dates: First submitted 2022-03-11; First posted 2022-04-08 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Bariatric Surgery Candidate; Weight Loss
Keywords: Bariatric surgery; Microbiota; Diet; Cognition; Brain structure
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples retained include serum, urine, plasma, stool for high-throughput sequencing of 16SrRNA and metagenomic shotgun sequencing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients undergoing bariatric surgery: Adult patients (≥ 30y yrs.) scheduled to undergo a first bariatric surgery recruited from the bariatric surgery clinic at the CIUSSS du Nord-de-l'Île-de-Montréal [N=120]
- Patients on the bariatric surgery waitlist: Age-, sex-, and BMI-matched waitlist control group [awaiting for bariatric surgery] recruited from the bariatric surgery clinic at the CIUSSS du Nord-de-l'Île-de-Montréal [N=60]
- Non-bariatric eligible individuals: Age-and sex-matched individuals who are not eligible for bariatric surgery, as an additional non-bariatric comparison group [N=60]
  *The 60 age-and sex-matched non-bariatric participants will have data captured just once [at baseline] on a limited number of key assessments

SUMMARY:
Emerging evidence suggests that dietary and metabolic interventions could potentially target prevention and supportive therapies as well as treatments that may slow the clinical deterioration of neurodegenerative disorders. Though certain dietary patterns can impair specific cognitive domains, e.g., declines in reasoning and global cognition, there is still no consensus on the optimal diet to maintain brain health. Studies have also shown an association between the gut microbiome and neurocognition, as the microbiota can affect neuronal function through neurotransmitters and neuroactive microbial metabolites. Furthermore, studies indicate that diet may strongly influence the gut microbiota. However, the mechanisms for these complex relationships are still poorly understood. Bariatric procedures [i.e., weight loss surgeries] create a unique environment, in which a fast change in gut microbiota composition and dietary patterns occurs through surgery-induced intestinal and metabolic modifications, leading to changes in gut-brain communication. Interestingly, improvements in neurocognitive domains including memory and executive function have been reported post-bariatric surgery. However, there is large variability in these outcomes, indicating that the benefits are not universal. The goal of the current study is to explore the associations between dietary patterns and gut microbiota with cognition and brain structure, using bariatric surgery as an efficient naturalistic experimental design. This project will also explore potential mediators of diet-microbiome alterations as they relate to improvements in brain function and structure. A total of 120 adult patients (> 30y yrs.) scheduled to undergo a first bariatric surgery along with 60 age-, sex-, and BMI-matched waitlist control group will be recruited from the bariatric surgery clinic at the CIUSSS du Nord-de-l'Île-de-Montréal. These individuals will undergo assessments 3 months before surgery, as well as 6- and 12-months post-surgery, or an equivalent time for those on the waitlist. This study will also include 60 age-and sex-matched individuals who are not eligible for bariatric surgery as an additional healthy Canadian comparison group (only one assessment time point). Assessments taken during the data collection period will include: self-report information [e.g., sociodemographic and background information, health and diet behaviours]; information from medical records [e.g., medications usage, peri- and post-surgical complications, etc.]; physiological measures [i.e., blood, urine and fecal samples collection]; cognitive assessment [i.e., neuropsychological tests battery]; and brain imaging [i.e., structural MRI]. Collectively, this study is designed to provide critical information about potential individually targeted diet-based preventative strategies to reduce the development and progression of neurodegenerative disorders. Moreover, this project will explore potential mediators of diet-microbiome alterations as they relate to improvements in brain function and structure, and as such, it will provide essential information on key mechanisms, stimulating further research and the creation of parallel non-dietary therapeutic options.

DETAILED DESCRIPTION:
Dietary patterns are associated with cognitive function and brain morphology. Though certain dietary patterns can impair specific cognitive domains, e.g., declines in reasoning and global cognition, there is still no consensus on the optimal 'brain diet'. Studies have also shown an association between the gut microbiome and neurocognition. The microbiota can affect neuronal function through neurotransmitters and neuroactive microbial metabolites. Furthermore, studies indicate that diet may strongly influence the gut microbiota, likely via intestinal permeability and inflammation. However, the mechanisms for this complex relationship between diet, gut microbiome and cognition are still poorly understood. Most of the work to date has focused on the negative effects of a Western style diet, with its subsequent microbiota alterations leading to cognitive impairment, via reduced barrier integrity, increased neuroinflammation, and impaired insulin signaling. However, very little is known about positive dietary-microbiome interactions, especially in humans. Bariatric surgery is considered the most effective treatment for severe obesity and it's related comorbidities, with the Sleeve gastrectomy (SG) being the most commonly performed procedures worldwide. These procedures create a unique environment, in which a fast change in gut microbiota composition occurs through surgery-induced intestinal and metabolic modifications, leading to changes in gut-brain communication. Moreover, these same post-surgical alterations to the gastrointestinal tract are accompanied by profound changes in dietary patterns that, in turn, influence microbiota composition. Following bariatric surgery, dietary intake is altered both in quantity and quality; however, considerable individual variations in surgically-induced dietary patterns have been previously demonstrated. Interestingly, improvements in neurocognitive domains including memory and executive function have been reported post-bariatric surgery. However, there is large variability in these outcomes, indicating that the benefits are not universal. Additionally, the extant literature is limited by a small number of studies, meaning that the underling mechanisms remain unclear. Importantly, how bariatric surgery-induced modifications in both dietary patterns and the gut microbiome effect cognitive function have yet to be explored. Finally, the overall changes in the gut microbiome and diet post-surgery may enhance biological pathways (e.g., gut hormones, inflammation, and neuroactive metabolites) which can affect brain function and structure, but the nature of these changes have not been studied extensively. The EMBRACE trial (Evaluation the impact of radical nutrition and Microbiome changes on BRAin funCtion and structurE) is a prospective, 15-month longitudinal study that aims to elucidate the associations between dietary patterns and gut microbiota with cognition and brain structure, using an efficient naturalistic experimental design which causes major disruptions to both diet and the microbiome, i.e., bariatric surgery. The main goal of this study is to evaluate how changes in gut microbiota composition and dietary patterns from pre- to post-bariatric surgery are linked to improved cognition and brain structure over the medium-term (12-months post-surgery). This project also aims to explore the potential mediating biological (e.g., inflammatory markers, hormonal changes, altered micronutrients levels and neuroactive microbial metabolites) pathways which might explain these relationships.

Primary aim: To evaluate the effect of surgery-induced changes in gut microbiota composition and dietary patterns from 3-M pre-surgery to 6-M post-surgery on 12-M post-surgical cognition, measured using sensitive neuropsychological tests.

Secondary aim: To evaluate the effect of surgery-induced changes in gut microbiota composition and dietary patterns from 3-M pre-surgery to 6-M post-surgery on 12-M post-surgical brain structure measured with magnetic resonance imaging (MRI) to assess brain volume, white-matter hyperintensities and cortical thickness.

Hypotheses for aims 1 and 2: Better quality microbiota and diet clusters (e.g., increased bacterial richness and diversity and greater low-saturated fat/high fibre intake) will be associated with increased performance on cognitive measures (higher total score on the neuropsychological test battery [primary] and its subscales [secondary]) and positive changes in brain measures (regional brain volume, hippocampal volume, cortical thickness and white-matter hyperintensities).

Exploratory aim: To examine biological changes (e.g., inflammatory state, hormonal changes, altered micronutrients levels and neuroactive microbial metabolites) pre- to post-surgery as potential mediating factors between microbiota/diet changes and cognitive/brain measures. Outcome: We will explore what post-surgical biological measures (e.g., reduced inflammatory markers, lower leptin levels, etc.) might mediate or moderate the links between specific microbiota and diet clusters and changes in cognitive function and brain measures.

A total of 120 adult patients (≥ 30y yrs.) scheduled to undergo a first bariatric surgery along with 60 age-, sex-, and BMI-matched waitlist control group will be recruited and undergo assessments 3 months before surgery, as well as 6- and 12-months post-surgery, or an equivalent time for those on the waitlist. This study will also include the recruitment of 60 age-and sex-matched individuals who are not eligible for bariatric surgery, as an additional non-bariatric comparison group. Evaluations will include standardized questionnaires on demographics, health behaviors and eating habits, physiological assessments (anthropometrics, inflammatory and blood-based measurements, 24-hour urine and fecal sample collection), cognitive assessment by neuropsychological tests, and structural magnetic resonance imaging (MRI).

Cluster analyses of the dietary and microbial alterations will define the various dietary patterns and microbiome profiles, then using repeated-measures mixed models, their associations with global cognitive changes and structural brain alterations will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 years or older
* Indeviduals planning to be available for two years of follow-up
* Ability ro read and speak French or English

Exclusion Criteria:

* A previous bariatric surgery
* Using long-term antibiotics
* Using commercially available prebiotic/probiotic in the past month
* A history of significant intestinal disease/disorder that would influence the microbiome (e.g., Crohn's disease)
* A non-bariatric surgery in the 6 months before being recruited
* A diagnosed neurologic disorder or deficits (e.g., dementia, stroke, or seizures)
* A diagnosis of a severe axis 1 psychotic disorder (e.g., schizophrenia) or bipolar disorder
* A current infection or a diagnosed infectious disease
* Pregnacy or breast feeding
* Active cancer
* Advanced kidney disease
* Advanced liver disease
* Past organ transplantation
* Having any contraindications for undergoing MRI [i.e., having a cardiac pacemaker (or pacemaker), defibrillator (a heart rhythm device), heart valve prosthesis (a prosthesis in the heart), Swan-Ganz catheter (a tube in the pulmonary artery on the chest), metal insulin or chemotherapy pump under the skin, neurostimulator, brain aneurysm clip (a clip in a blood vessel of the brain), metal prosthesis or rods (following surgery), metal cerclage (metal support on a bone), cochlear or ocular implant (an implant in the ear or eye), penile implant, an intraocular metal fragment (metal debris in the eye), an intrauterine device that does not conform with the MRI, any plastic implants (e.g., breasts) or a patch on the skin for the administration of a medication unless it can remove before scan session]. Additional requirements for MRI includes patients agreement to: 1) have a pregnancy test and remove makeup, 2) the removal of dentures (full or partial), and 3) provide information on all surgery and previous tattoos (tattoos made for many years or those made in some countries, as the ink contains metallic particles).
* For participants included in the non-bariatric eligible comparison group group, individuals with any physician diagnosed major non-communicable chronic disease, defined as cardiovascular disease, chronic obstructive lung disease, cancer, diabetes, or obesity, will be excluded.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 120 adult patients (≥ 30y yrs.) scheduled to undergo a first bariatric surgery (i.e., no previous surgery-related disruption to the gut microbiota), along with 60 age-, sex-, and BMI-matched waitlist control group will be recruited from the bariatric surgery clinic at the CIUSSS du Nord-de-l'Île-de-Montréal, which conducts around 1,000 surgeries per year with a waitlist of approximately 1,000 individuals, with an average wait of 3 years.
  Volunteers for the non-bariatric eligible individuals group [healthy control group] will be recruited using advertisements, recruitment materials will include a short description of the study and details of who is eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Changes in cognition from baseline [3 months pre-surgery] to 12 months post-surgery, measured using sensitive neuropsychological test battery [NTB] | 3 months pre- and 12 months post-surgery [or equivalent time point for waitlist participants]
  Global cognition will be assessed using the NTB total score (the primary outcome), a composite NTB score of 14 sub-tests. NTB domain Z scores for executive functioning, processing speed, and memory will also be calculated.

SECONDARY OUTCOMES:
Changes in MRI-derived brain volume from baseline [3 months pre-surgery] to 12 months | 3 months pre- and 12 months post-surgery [or equivalent time point for waitlist participants]
  Participants will be scanned on a Siemens 3T Prisma Fit MRI system (Siemens Medical Solutions, Erlangen, Germany). The MRI protocol will use structural sequences of the CIMAQ/Canadian Dementia Imaging Protocol (www.cdip-pcid.ca). The session contains a 3D T1-weighted MRI for volumetric and cortical thickness analyses (TR/TE 2300/2.98 ms; 9° flip angle; voxel size: 1x1x1 mm).
Changes in MRI-derived white-matter hyperintensities from baseline [3 months pre-surgery] to 12 months post-surgery | 3 months pre- and 12 months post-surgery [or equivalent time point for waitlist participants]
  Participants will be scanned on a Siemens 3T Prisma Fit MRI system (Siemens Medical Solutions, Erlangen, Germany). The MRI protocol will use structural sequences of the CIMAQ/Canadian Dementia Imaging Protocol (www.cdip-pcid.ca). The session contains FLAIR sequences (TR/TE 9000/129 ms; voxel size: 1×1×1 mm, for white matter hyperinsities (WMH) analyses.

OTHER OUTCOMES:
Trajectories of clusters of gut microbiota composition measured with Metagenomic shotgun sequencing from baseline through to 12 months post-surgery | 3 months pre- and 6 and 12 months post-surgery [or equivalent time point for waitlist participants]
  Whole genomes will be sequenced using Illumina paired-end 150bp sequencing to achieve 20-30Gb sequences per sample. Microbiome changes at the levels of the community (richness, diversity), taxa including absolute and relative abundance of microbes classified along the different levels of the tree of life (family, genera, species), and functions (genes and pathways abundances) will be evaluated by metagenomic tools (i.e., R/Bioconductor packages such as vegan, phyloseq, microbiome, and MaAslin2).
Trajectories of clusters of gut microbiota composition measured with High-throughput sequencing of 16 S rRNA genes from baseline through to 12 months post-surgery | 3 months pre- and 6 and 12 months post-surgery [or equivalent time point for waitlist participants]
  Resulting sequences will be clustered into operational taxonomic units (OTUs) by applying a cut-off of 97% similarity using the Greengenes reference database. Alpha-diversity metrics, Shannon [species evenness and diversity]) will be calculated from the rarefied OTUs. The β-diversity will be estimated using UniFrac and Bray-Curtis distances and visualized using principal coordinate analysis (PCoA).
Trajectories of macro-level dietary intake from baseline through to 12 months post-surgery | 3 months pre- and 6 and 12 months post-surgery [or equivalent time point for waitlist participants]
  A 7-day food diary with photo capture via a mobile application (Keenoa), will be used to collect dietary data. Data from the food diaries will be analyzed using the Canadian Nutrient File, a Government of Canada food database.
Trajectories of diet quality measured by the Healthy Eating Index (HEI) from baseline through to 12 months post-surgery | 3 months pre- and 6 and 12 months post-surgery [or equivalent time point for waitlist participants]
  The Healthy Eating Index (HEI) will be used as an index of overall diet quality, specifically for a Canadian population. An ideal overall HEI score of 100 reflects that the set of foods aligns with key dietary recommendations from the Dietary Guidelines for Canadians.
Trajectories of dietary inflammatory Index from baseline through to 12 months post-surgery | 3 months pre- and 6 and 12 months post-surgery [or equivalent time point for waitlist participants]
  The Dietary inflammatory Index [DII] measure the potential impact of a diet on an individual's inflammatory status, and it has been validated mainly in Western countries. A high DII score reflects pro-inflammatory potential of the diet, whereas a low DII score reflects the anti-inflammatory potential of the diet
Trajectories of mediterranean diet adherence from baseline through to 12 months post-surgery | 3 months pre- and 6 and 12 months post-surgery [or equivalent time point for waitlist participants]
  The Mediterranean Diet Adherence Screener (MEDAS) is a 14-item instrument that enables a rapid assessment of adherence to the Mediterranean diet. The final MEDAS score can range between 0 and 14, higher scores reflects higher level of adherence to the mediterranean diet.
Trajectories of food tolerance from baseline through to12 months post-surgery | 3 months pre- and 6 and 12 months post-surgery [or equivalent time point for waitlist participants]
  Food tolerance after bariatric surgery will be assessed by the validated, self-reported questionnaire for quick assessment of food tolerance after bariatric surgery with a score of 1 to 27. This instrument consists of 4 components, including overall patient satisfaction with alimentation, the timing and content of meals and snacks, the tolerance of different types of foods, and the frequency of vomiting. Higher scores reflects higher level of tolerance to food and eating post-surgery.
Trajectories of Eating behavior from baseline through to 12 months post-surgery | 3 months pre- and 6 and 12 months post-surgery [or equivalent time point for waitlist participants]
  The Dutch Eating Behavior Questionnaire (DEBQ) evaluates emotional eating behaviors, external eating behaviors, and restricted eating behaviors, and is composed of 33 items, that are evaluated by a 5-point Likert scale (one: never, two: rarely, three: sometimes, four: often, and five: very often). Items on the subscales are averaged, with higher mean scores indicative of greater restrained eating, eating in response to emotions, and eating triggered by external cues.
Trajectories of binge eating from baseline through to 12 months post-surgery | 3 months pre- and 6 and 12 months post-surgery [or equivalent time point for waitlist participants]
  The Binge-Eating Disorder Screener (BEDS-7) will be used to identify individuals with probable binge-eating disorder (BED). This is a brief, patient-reported screening tool designed to identify individuals with probable binge-eating disorder (BED).
Trajectories of eating self-efficacy from baseline through to 12 months post-surgery | 3 months pre- and 6 and 12 months post-surgery [or equivalent time point for waitlist participants]
  The Weight Efficacy Lifestyle Questionnaire (WEL) is a commonly used measure of eating self-efficacy consisting of 20-items and five situational factors. Higher WEL scores indicate higher self-efficacy to resist eating.
Trajectories of grazing eating behavior from baseline through to 12 months post-surgery | 3 months pre- and 6 and 12 months post-surgery [or equivalent time point for waitlist participants]
  The grazing questionnaire will be used, this instrument include seven-item self-report scale measuring the frequency of unplanned, continuous and repetitive eating of small amounts of food [i.e., grazing eating behavior].
Trajectories of excess weight loss from baseline through to 12 months post-surgery | 3 months pre- and 6 and 12 months post-surgery [or equivalent time point for waitlist participants]
  Weight will be measured on a digital medical scale; height will be measured by a stadiometer and BMI will be calculated by weight divided by the height squared. Percentages of excess weight loss (% EWL) will be calculated as follows: [(preoperative weight-postoperative weight)/ (preoperative weight - ideal weight)] × 100. Ideal body weight (IBW) will be considered the weight for a BMI 25 kg/m2.
Trajectories of urine nitrogen as a biomarker for dietary protein intake, from baseline through to 12 months post-surgery | 3 months pre- and 6 and 12 months post-surgery [or equivalent time point for waitlist participants]
  Dietary 24-hour urinary biomarkers measured for objective verification for some of the self-reported food intakes will include urine Nitrogen that will be used as a biomarker for the validation of dietary protein intake. 24-hour urine collection will be performed by participants following each lab visit with the full instructions given by a research assistant at each lab visit.
Trajectories of urine Alkylresorcinols (ARs) and their metabolites as a biomarker for fiber and whole grain products intake, from baseline through to 12 months post-surgery | 3 months pre- and 6 and 12 months post-surgery [or equivalent time point for waitlist participants]
  Dietary 24-hour urinary biomarkers measured for objective verification for some of the self-reported food intakes will include Alkylresorcinols (ARs) and their metabolites (3-(3,5-dihydroxyphenyl)-propanoic acid (DHPPA) and 3,5-dihydroxybenzoic acid (DHBA)) that will be used as markers for fiber and whole grain products.
Trajectories of urine fructose as a biomarkers for sugar intake from baseline through to 12 months post-surgery | 3 months pre- and 6 and 12 months post-surgery [or equivalent time point for waitlist participants]
  Fructose 24 hours urine excretion will be used to assess added, natural, and total sugar intake.
Trajectories of urine sodium as a biomarkers for total sodium intake from baseline at 6 through to 12 months post-surgery | 3 months pre- and 6 and 12 months post-surgery [or equivalent time point for waitlist participants]
  Sodium and albumin 24 hour excretions will be used to assess sodium intake.
Trajectories of urine potassium as a biomarkers for total potassium intake from baseline through to 12 months post-surgery | 3 months pre- and 6 and 12 months post-surgery [or equivalent time point for waitlist participants]
  Potassium 24 hour excretions will be used to assess potassium intake.
Trajectories of Quality of Life from baseline through to 12 months post-surgery | 3 months pre- and 6 and 12 months post-surgery [or equivalent time point for waitlist participants]
  The European Quality of Life Five Dimensions Questionnaire [EQ-5D] is a standardized measure that will be used to collect data about participant's quality of life, and have been previously used within Quebec population.
Trajectories of depressive symptoms from baseline through to 12 months post-surgery | 3 months pre- and 6 and 12 months post-surgery [or equivalent time point for waitlist participants]
  The Beck Depression Inventory-II (BDI-II), a 21-item questionnaire self-report measure will be used to assess depressive symptomatology. Sum scores ranging from zero to 13 indicate minimal depression, 14 to 19 indicate mild depression, 20 to 28 indicate moderate depression, and 29 to 63 indicate severe depression.
Trajectories of physical activity from baseline through to 12 months post-surgery | 3 months pre- and 6 and 12 months post-surgery [or equivalent time point for waitlist participants]
  Physical activity information will be collected using the Godin Leisure-Time Exercise Questionnaire.
  Alcohol consumption and smoking behaviour will be assessed using questions adapted from Statistics Canada's alcohol and other drugs survey. The usage of nutritional and vitamin supplements will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Bacon, PhD, Principal Investigator — Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Locations (1):
- Hopital du Sacre-Coeur de Montreal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No